CLINICAL TRIAL: NCT04190745
Title: Zhejiang Cancer Hospital
Brief Title: Toripalimab Combined With Apatinib Mesylate for the Treatment of Gastric Adenocarcinoma in a Prospective Randomized Multicenter Phase II Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2019-155
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Experimental)
  Interventions: Drug: paclitaxel
- The experimental group (Experimental)
  Interventions: Drug: Toripalimab+Apatinib mesylate

INTERVENTIONS:
Drug: Toripalimab+Apatinib mesylate — Toripalimab 240mg, ivgtt, Q3w Apatinib mesylate 250mg PO. QD
  Arms: The experimental group
Drug: paclitaxel — paclitaxel 80mg/m2, q3w
  Arms: The control group

SUMMARY:
Preclinical studies have shown that Toripalimab and Nivolumab and Pembrolizumab have similar safety but better in vivo efficacy than target monoclonal antibody candidates with different sequence characteristics.In addition, apatinib mesylate is a small-molecule drug that can target VEGFR and is itself a powerful therapeutic drug for gastric cancer, so we designed a clinical trial of apatinib combined with toripalimab monoclonal antibody.The study focused on 12 month OS rate, progression-free survival (PFS), clinical objective response rate (ORR), and drug safety.The study was an open, multicenter, randomized controlled clinical trial with a 1:1 distribution of trial and control groups.It is expected that 58 people will be included in the experimental group and 58 people in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Have fully understood the study and voluntarily signed the informed consent (ICF);
* Pathologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma, except siwert I type;
* Previously received an anti-tumor drug therapy for advanced gastric adenocarcinoma and identified tumor progression or intolerance to existing chemotherapy regimens; If the radical surgery accompanied by adjuvant or neoadjuvant chemotherapy recurred or metastasized within 6 months after the end of the study, the patients could be enrolled in this study.
* At least one measurable lesion (according to RECIST 1.1);
* Agree to provide previously stored tumor tissue specimens or biopsy to collect tumor lesion tissues and send them to the central laboratory for pd-l1 IHC test;
* Age from 18 to 75, regardless of gender;
* ECOG score 0-1;
* Expected survival time ≥3 months;
* The laboratory inspection value must meet the following criteria within 7 days prior to enrollment:

  1. neutrophils ≥1.5×109/L;
  2. platelet ≥75×109/L;
  3. hemoglobin ≥90g/L (no infusion of concentrated red blood cells within 2 weeks);
  4. serum creatinine ≤1.5× the upper normal ULN, or creatinine clearance >50 mL/min;
  5. serum total bilirubin ≤1.5×ULN (subjects with gilbert syndrome are allowed to have total bilirubin ≤3×ULN);
  6. AST and ALT ≤2.5×ULN;For subjects with liver metastasis, ALT and AST≤5×ULN;
* Within 28 days before enrollment, women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraception during study drug use and within 60 days after the last dose. In this program, women of childbearing age are defined as sexually mature women: 1) women who have not undergone hysterectomy or bilateral ovariectomies; 2) women who have not experienced continuous natural menopause for 24 months (amenorrhea does not exclude fertility after cancer treatment) (i.e.* female spouses of male subjects should also follow the above contraceptive requirements if they are of childbearing age.

Exclusion Criteria:

* Those who are known to be allergic to the components of the experimental drug;
* Received anti-tumor cytotoxic drug therapy, biological drug therapy (such as monoclonal antibody), immunotherapy (such as interleukin-2 or interferon), or other study drug therapy within the first 4 weeks of enrollment;
* Received tyrosine kinase inhibitor treatment within 2 weeks before enrollment;
* Received radiotherapy within 4 weeks before enrollment, or received radiotherapy with radioactive drugs within 8 weeks, except local palliative radiotherapy for bone metastasis;
* Major surgery was performed or not fully recovered from the previous surgery within the first 4 weeks of enrollment (the definition of major surgery refers to the level 3 and level 4 surgery as stipulated in the administrative measures for clinical application of medical technology implemented on May 1, 2009);
* The toxicity of previous anti-tumor therapy has not recovered to CTCAE grade 0-1, except the following:

  1. loss of hair;
  2. pigmentation;
  3. peripheral neurotoxicity has been restored to <CTCAE level 2;
  4. Long-term toxicity caused by radiotherapy cannot be recovered according to the judgment of the researcher;
* Subjects with clinical symptoms of central nervous system metastasis (such as brain edema, need for hormone intervention, or progression of brain metastasis) or cancerous meningitis.Subjects who have received previous brain or meningeal metastasis treatment, if clinical stability has been maintained for at least 2 months, and who have stopped systemic sex hormone therapy (>10mg/ day prednisone or other effective hormones) for more than 4 weeks can be included;
* Previous or present coexisting malignancies (except well-controlled basal cell carcinoma of the skin, breast/cervical carcinoma in situ, and other well-controlled malignancies that have not been treated in the past five years);
* The subject has any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, hyperthyroidism and hypothyroidism;Subjects with vitiligo or asthma that had been completely relieved in childhood and who did not need any intervention in adulthood were included.Asthma that requires a bronchodilator for medical intervention is not included);
* Previous use of anti-pd-1 antibody, anti-pd-l1 antibody, anti-pd-l2 antibody or anti-ctla-4 antibody (or any other antibody acting on the T cell synergistic stimulation or checkpoint pathway);
* Her2+ positive patients who had not received trastuzumab treatment in the past
* Subjects with active tuberculosis (TB) were receiving anti-tb treatment or had received anti-tb treatment within 1 year before screening;
* Comorbiditis requiring long-term use of immunosuppressive drugs or systemic or local use of corticosteroids with immunosuppressive doses (>10mg/d prednisone or other therapeutic hormones);
* Received any anti-infection vaccine (such as influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before enrollment;
* pregnant or lactating women;
* HIV positive;
* HBsAg positive and HBV DNA copy number positive (quantitative detection ≥1000cps/ml);
* Positive blood screening for chronic Hepatitis c (HCV antibody positive);
* Any other disease or condition of clinical significance that the investigator considers may affect protocol compliance or the subject's signing of an informed consent form (ICF), or is not appropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Subjects' Overall survival rate at 12 months | 12 months
  Overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Jieer Ying, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei Q, Xu X, Li J, Wang C, Chen W, Xie Y, Luo C, Chen L, Chu J, Wu W, Han Z, Yang Y, Hu Z, Xu Q, Ying J. Apatinib Plus Toripalimab (Anti-PD1 Therapy) as Second-Line Therapy in Patients With Advanced Gastric or Esophagogastric Junction Cancer: Results From a Randomized, Open-Label Phase II Study. Oncologist. 2024 Apr 4;29(4):364-e578. doi: 10.1093/oncolo/oyae005. PMID 38366886